CLINICAL TRIAL: NCT02527122
Title: Dermatophagoides Pteronyssinus and Dermatophagoides Farinae Allergen Extract. Determination of the Allergenic Potency in Vivo Histamine Equivalent Units (HEP)
Brief Title: Biological Stardadization of D. Pteronyssinus and D. Farinae Allergen Extracts
Acronym: MM09
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MM09-STD-011; 2013-005394-45 (EudraCT Number)
Record Dates: First submitted 2015-08-17; First posted 2015-08-18 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Immune System Diseases
Keywords: Immune System Diseases; Prick Test; Dermatophagoides pteronyssinus; Dermatophagoides farinae
MeSH Terms: conditions — Immune System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allergen extracts (Experimental): Skin prick test of 4 concentrations of D. pteronyssinus allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of one forearm. Assessment of the wheal size after 15 minutes.
  Skin prick test of 4 concentrations of D. farinae allergen extract, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the other forearm. Assessment of the wheal size after 15 minutes.
  Interventions: Diagnostic Test: Allergen extracts

INTERVENTIONS:
Diagnostic Test: Allergen extracts

SUMMARY:
Four concentrations of Dermatophagoides pteronyssinus and Dermatophagoides farinae allergen extracts, together with a positive and negative control, using 10 mg/ml histamine dihydrochloride solution and a glycerinated phenol saline solution, respectively, will be tested in every patient in duplicate on the volar surface of the forearm..

DETAILED DESCRIPTION:
This is an open, unblinded and non-randomized biological assay. The study design is a slight modification of the recommendations proposed by the Nordic Guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Clinical history positive inhalation allergy (rhinitis I rhinoconjunctivitis I asthma) against Dermatophagoides pteronyssinus or Dermatophagoides farinae.
* A prick-test positive (average of the papule ≥ 3 mm diameter) with a summary of the same allergen I presence against the allergen specific Immunoglobulin E.
* The average area of the papule obtained by histamine dihydrochloride to 10 mgml must be greater than or equal 7 mm2.
* Age: over 18 years of age.
* Both sexes.

Exclusion Criteria:

* Subjects outside of the age range.
* Individuals who have previously received immunotherapy in the last 5 years for the treatment of asthma or the allergic rhinoconjunctivitis induced by allergens that may interfere with the extract mixture of Dermatophagoides pteronyssinus or farinae.
* Subjects with important symptoms of rhinoconjunctivitis I bronchial asthma in which the suspension of the antihistamine treatment for systemic is contraindicated.
* Subjects that have previously submitted a serious secondary reaction during skin prick test diagnostic tests.
* Subjects in treatment with ss-blockers.
* Unstable subjects of clinical point of view (asthma acute, febrile, etc.).
* Subjects with lesions of active hives, severe active dermographism, severe atopic dermatitis, sunburn, eczema, lesions of psoriasis in the area of realization of the prick test (risk of false positives).
* Subjects with viral infection activates the herpes simplex or herpes varicella-zoster in the area of realization of the prick test.
* Subjects that have some pathology in which the administration of adrenaline (hyperthyroidism, hypertension, heart disease, etc.) is contraindicated.
* States of the subject that can not offer cooperation and severe psychiatric disorders.
* Pregnant or women at risk of pregnancy and breastfeeding women.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
The wheal size diameter on the skin at the site of the puncture during the immediate phase when applied each concentration of the allergen extract | 1 hour
  wheal size diameter OF THE SKIN PRICK TEST

CONTACTS AND LOCATIONS:
Overall Officials: Elena Rodríguez, MD, Study Director
Locations (1):
- Hospital Univ. Ntra. Sra. de la Candelaria, Santa Cruz de Tenerife, Canary Islands, Spain

IPD SHARING:
Plan to Share IPD: No